CLINICAL TRIAL: NCT04319276
Title: A Phase 1 Clinical Trial of Oral Gallium Maltolate for the Treatment of Relapsed and Refractory Glioblastoma
Brief Title: Oral Gallium Maltolate for the Treatment of Relapsed and Refractory Glioblastoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Jennifer Connelly, MD, Professor, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRO00041263
Record Dates: First submitted 2020-03-20; First posted 2020-03-24 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Glioblastoma
Keywords: gallium maltolate; Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — gallium maltolate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Dose-escalation Phase (500 mg) (Experimental): This is a 3 + 3 design. Participants will be entered sequentially. If 0 of 3 participants has a dose-limiting toxicity (DLT), new participants may be entered at the next higher dose level. If 1 of 3 participants has a DLT, up to 3 more participants are to be treated at that same dose level. If 0 of the additional 3 participants at that dose level has a DLT, new participants may be entered at the next higher dose level. If 1 or more of the additional 3 participants experience a DLT, 0 participants are to be started at that dose level and the preceding dose is the maximum-tolerated dose (MTD). If 2 of 3 of the dosed participants has a DLT on the first dose level, the drug will be administered at a lower dose. If 0 of 3 participants has a DLT at the highest dose level, an additional 3 participants will be enrolled to ensure that 6 participants are treated at the MTD. The MTD is the highest dose level at which no more than 1 of 6 treated participants, experiences a DLT.
  Interventions: Drug: Gallium maltolate (500 mg)
- Dose-escalation Phase (1,000 mg) (Experimental): This is a 3 + 3 design. Participants will be entered sequentially. If 0 of 3 participants has a dose-limiting toxicity (DLT), new participants may be entered at the next higher dose level. If 1 of 3 participants has a DLT, up to 3 more participants are to be treated at that same dose level. If 0 of the additional 3 participants at that dose level has a DLT, new participants may be entered at the next higher dose level. If 1 or more of the additional 3 participants experience a DLT, 0 participants are to be started at that dose level and the preceding dose is the maximum-tolerated dose (MTD). If 2 of 3 of the dosed participants has a DLT on the first dose level, the drug will be administered at a lower dose. If 0 of 3 participants has a DLT at the highest dose level, an additional 3 participants will be enrolled to ensure that 6 participants are treated at the MTD. The MTD is the highest dose level at which no more than 1 of 6 treated participants, experiences a DLT.
  Interventions: Drug: Gallium maltolate (1,000 mg)
- Dose-escalation Phase (1,500 mg) (Experimental): This is a 3 + 3 design. Participants will be entered sequentially. If 0 of 3 participants has a dose-limiting toxicity (DLT), new participants may be entered at the next higher dose level. If 1 of 3 participants has a DLT, up to 3 more participants are to be treated at that same dose level. If 0 of the additional 3 participants at that dose level has a DLT, new participants may be entered at the next higher dose level. If 1 or more of the additional 3 participants experience a DLT, 0 participants are to be started at that dose level and the preceding dose is the maximum-tolerated dose (MTD). If 2 of 3 of the dosed participants has a DLT on the first dose level, the drug will be administered at a lower dose. If 0 of 3 participants has a DLT at the highest dose level, an additional 3 participants will be enrolled to ensure that 6 participants are treated at the MTD. The MTD is the highest dose level at which no more than 1 of 6 treated participants, experiences a DLT.
  Interventions: Drug: Gallium maltolate (1,500 mg)
- Dose-escalation Phase (2,000 mg) (Experimental): This is a 3 + 3 design. Participants will be entered sequentially. If 0 of 3 participants has a dose-limiting toxicity (DLT), new participants may be entered at the next higher dose level. If 1 of 3 participants has a DLT, up to 3 more participants are to be treated at that same dose level. If 0 of the additional 3 participants at that dose level has a DLT, new participants may be entered at the next higher dose level. If 1 or more of the additional 3 participants experience a DLT, 0 participants are to be started at that dose level and the preceding dose is the maximum-tolerated dose (MTD). If 2 of 3 of the dosed participants has a DLT on the first dose level, the drug will be administered at a lower dose. If 0 of 3 participants has a DLT at the highest dose level, an additional 3 participants will be enrolled to ensure that 6 participants are treated at the MTD. The MTD is the highest dose level at which no more than 1 of 6 treated participants, experiences a DLT.
  Interventions: Drug: Gallium maltolate (2,000 mg)
- Dose-escalation Phase (2,500 mg) (Experimental): This is a 3 + 3 design. Participants will be entered sequentially. If 0 of 3 participants has a dose-limiting toxicity (DLT), new participants may be entered at the next higher dose level. If 1 of 3 participants has a DLT, up to 3 more participants are to be treated at that same dose level. If 0 of the additional 3 participants at that dose level has a DLT, new participants may be entered at the next higher dose level. If 1 or more of the additional 3 participants experience a DLT, 0 participants are to be started at that dose level and the preceding dose is the maximum-tolerated dose (MTD). If 2 of 3 of the dosed participants has a DLT on the first dose level, the drug will be administered at a lower dose. If 0 of 3 participants has a DLT at the highest dose level, an additional 3 participants will be enrolled to ensure that 6 participants are treated at the MTD. The MTD is the highest dose level at which no more than 1 of 6 treated participants, experiences a DLT.
  Interventions: Drug: Gallium maltolate (2,500 mg)
- Dose-expansion Phase (Experimental): A minimum of six participants will be enrolled in the dose expansion phase for a total of 12 subjects at the recommended phase 2 dose.
  Interventions: Drug: Gallium maltolate (recommended phase 2 dose)

INTERVENTIONS:
Drug: Gallium maltolate (500 mg) — This is a 3+3 design. The doses are as follows: level -1: 500 mg every other day; level 0: (starting dose) 500 mg daily; level 1: 1,000 mg daily; level 2: 1,500 mg daily; level 3: 2,000 mg daily; level 4: 2,500 mg daily.
  Other Names: Chemical Abstracts Service (CAS) 108560-70-9
  Arms: Dose-escalation Phase (500 mg)
Drug: Gallium maltolate (1,000 mg) — This is a 3+3 design. The doses are as follows: level -1: 500 mg every other day; level 0: (starting dose) 500 mg daily; level 1: 1,000 mg daily; level 2: 1,500 mg daily; level 3: 2,000 mg daily; level 4: 2,500 mg daily.
  Other Names: CAS 108560-70-9
  Arms: Dose-escalation Phase (1,000 mg)
Drug: Gallium maltolate (1,500 mg) — This is a 3+3 design. The doses are as follows: level -1: 500 mg every other day; level 0: (starting dose) 500 mg daily; level 1: 1,000 mg daily; level 2: 1,500 mg daily; level 3: 2,000 mg daily; level 4: 2,500 mg daily.
  Other Names: CAS 108560-70-9
  Arms: Dose-escalation Phase (1,500 mg)
Drug: Gallium maltolate (2,000 mg) — This is a 3+3 design. The doses are as follows: level -1: 500 mg every other day; level 0: (starting dose) 500 mg daily; level 1: 1,000 mg daily; level 2: 1,500 mg daily; level 3: 2,000 mg daily; level 4: 2,500 mg daily.
  Other Names: CAS 108560-70-9
  Arms: Dose-escalation Phase (2,000 mg)
Drug: Gallium maltolate (2,500 mg) — This is a 3+3 design. The doses are as follows: level -1: 500 mg every other day; level 0: (starting dose) 500 mg daily; level 1: 1,000 mg daily; level 2: 1,500 mg daily; level 3: 2,000 mg daily; level 4: 2,500 mg daily.
  Other Names: CAS 108560-70-9
  Arms: Dose-escalation Phase (2,500 mg)
Drug: Gallium maltolate (recommended phase 2 dose) — The maximum-tolerated dose (recommended phase 2 dose).
  Other Names: CAS 108560-70-9
  Arms: Dose-expansion Phase

SUMMARY:
This is a phase 1 investigational study to assess the safety and preliminary efficacy of oral gallium maltolate (GaM) in participants with relapsed glioblastoma (GBM).

DETAILED DESCRIPTION:
This is a prospective, single-center, single-arm, open-label phase 1 study to determine the antineoplastic activity, safety and tolerance of GaM in participants with relapsed, treatment-refractory GBM. Although GaM has been studied in previous phase 1 clinical trials in normal individuals and in participants with a variety of different solid tumors, it has never been evaluated in this population of participants. Dosages in this study have been defined to have limited side effects in other phase 1 trials. The maximum number of participants to enroll in the dose escalation part will not exceed 36. The trial will follow a 3 + 3 phase I dose escalation design.

ELIGIBILITY:
Inclusion Criteria

1. Voluntary written consent must be obtained before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
2. All patients must have a prior histological diagnosis of GBM (WHO grade IV) or molecular features of GBM (per the 6th volume of Central Nervous System Tumors in the 5th edition of the WHO Classification of Tumors).
3. Patients are required to have received standard treatment which consists of radiotherapy and temozolomide [i.e., the Stupp Protocol (3)] Treatment with adjuvant temozolimide must be completed at least four weeks prior to GaM administration to avoid potential for overlapping toxicity with GaM. Although the half-life (T½) of temozolomide is 1.8 hours and it would be expected to be cleared by five half-lives, some patients receiving temozolomide may experience a delayed suppression of their ANC. Hence, a four-week interval between completion of temozolomide and GaM will be required. There is no maximum limit to the amount of chemotherapy or radiation patients have received prior to enrollment.
4. Patients must have measurable disease that can be assessed for response to treatment as defined by the Response Assessment in Neuro-Oncology (RANO) criteria which incorporates MRI assessment and clinical factors. In the absence of measurable disease, pathologic confirmation of recurrent disease is required.
5. Male or female subjects must be ≥18 years of age.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
7. Patients must have adequate bone marrow function as evidenced by:

   1. an absolute neutrophil count (ANC) of >1500/μL (stable off any growth factor within one week of study drug administration
   2. Hemoglobin > 9 g/dL
   3. Platelet count > 100.000/μL without transfusion within one week
8. Patients must have adequate hepatic and renal function based on the following laboratory tests: a. alanine transaminase (ALT) ≤ 2 x upper limits of normal (ULN) b. aspartate aminotransferase (AST) ≤ 2 x ULN c. Alkaline phosphatase ≤ 2 x ULN d. Total bilirubin ≤ 2 x ULN e. Creatinine < 1.5 mg/dL or glomerular filtration rate (GFR) by Modification of Diet in Renal Disease (MDRD) > 45
9. Female subjects must meet one of the following:

   * Postmenopausal for at least one year before enrollment, OR
   * Surgically sterile (i.e., undergone a hysterectomy or bilateral oophorectomy), OR
   * If subject is of childbearing potential (defined as not satisfying either of the above two criteria), agree to practice two acceptable methods of contraception (combination methods require use of two of the following: diaphragm with spermicide, cervical cap with spermicide, contraceptive sponge, male or female condom, hormonal contraceptive) from the time of signing of the informed consent form through 21days after the last dose of study agent, OR
   * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable contraception methods.)
10. Male subjects, even if surgically sterilized (i.e., status post-vasectomy), must agree to one of the following:

    * Practice effective barrier contraception during the entire study period and through 60 calendar days after the last dose of study agent, OR
    * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)
11. Patients taking oral iron supplements or iron chelators must discontinue these medications at least one week prior to starting GaM since these agents may impact on the efficacy of GaM. Drug-drug interactions between GaM and other concomitant medications have not been reported.

Exclusion Criteria

1. Presence of other active malignant disease diagnosed within 12 months, with the exception of adequately treated non-melanoma skin cancer, adequately treated melanoma grade 2 or less, or cervical intraepithelial neoplasia. Active malignancy is malignancy receiving treatment.
2. Prior chemotherapy or radiotherapy within 14 days of study entry.
3. Known hypersensitivity to or intolerance to gallium-based medications.
4. Concurrent use of cytotoxic chemotherapy is not permitted.
5. Unstable or severe concurrent medical conditions such as severe heart (New York Heart Association Class 3 or 4) or known lung (FEV <50%) disease, uncontrolled diabetes mellitus.
6. History of interstitial lung disease, history of slowly progressive dyspnea and unproductive cough, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, pulmonary hypersensitivity pneumonitis, or symptomatic pleural effusion.
7. Patients who have not completed all standard-of-care treatments including surgical procedures and radiation therapy.
8. Inability to tolerate an oral medication or keep pills down.
9. Patients who are pregnant or nursing.
10. Patients with any condition which, in the investigator's opinion, makes the patient unsuitable for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2025-02-13 (Actual); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Maximum-tolerated dose. | Each 28-day cohort
  This will be determined from the incidence of dose limiting toxicities at each dosage.

SECONDARY OUTCOMES:
Progression-free survival | 6 months
  This measure is the number of months participants remain free from evidence of disease. Imaging will be done every eight weeks and reported at six months.
Overall survival | 6 months
  Overall survival is determined as the average number of months subjects survived following enrollment.
Dose-limiting toxicity | 28 days for each cohort
  Number of participants experiencing a dose limiting toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Connelly, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital & the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No